CLINICAL TRIAL: NCT01684241
Title: Clinical First-in-human Dose Escalation Study Evaluating the Safety and Tolerability of Intranodal Administration of an RNA-based Cancer Vaccine Targeting Two Tumor-associated Antigens in Patients With Advanced Melanoma
Brief Title: RBL001/RBL002 Phase I Clinical Trial
Acronym: MERIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech RNA Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB_0001-01
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Melanoma
Keywords: Biontech; Biontech RNA Pharmaceuticals GmbH; Biontech RNA; MERIT; RNA; Immuno Therapy; RB_0001-01; Ribological; Melanoma; RBL001; RBL002; cancer vaccine
MeSH Terms: conditions — Melanoma | interventions — Cancer Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RBL001/RBL002 intranodal administration (Experimental): All participants will be treated with RBL001/RBL002 after allocation to one of the four escalating dose cohorts:
  * Cohort-1 50 µg RBL001 and 50 µg RBL002
  * Cohort-2 100 µg RBL001 and 100 µg RBL002
  * Cohort-3 300 µg RBL001 and 300 µg RBL002
  * Cohort-4 600 µg RBL001 and 600 µg RBL002
  Interventions: Biological: RBL001/RBL002

INTERVENTIONS:
Biological: RBL001/RBL002 — Each participant will receive 8 repeated intranodal administrations of RBL001 and RBL002 during a time frame of 43 to 51 days.
  Other Names: cancer vaccine

SUMMARY:
Clinical first-in-human dose escalation study evaluating the safety and tolerability of intranodal administration of an RNA-based cancer vaccine targeting two tumor-associated antigens in patients with advanced melanoma

DETAILED DESCRIPTION:
RBL001/RBL002 are naked ribonucleic acid (RNA) based recombinant vaccines that were optimized to induce antigen specific CD8+ and CD4+ T cell responses against malignant melanoma target antigens.

The Targeted antigens are well characterized antigens in melanoma that have been previously utilized with excellent safety and proven immunogenicity as vaccine targets in a number of independent clinical trials.

The overall rationale of the study is to determine safety of the novel RNA based vaccine approach and determine vaccine target antigen directed immune responses as early biomarkers for clinical mode of action.

The RBL001/RBL002 vaccine is expected to lead to several effects contributing to its immunological (therapeutic) effect. First, ultrasound guided administration of naked RNA drug product into lymph nodes is expected to result in rapid uptake of naked RNA by lymph node resident professional antigen-presenting cells (APCs). Incorporated RNA is known to translocate to the cytoplasm leading to its translation by the host ribosome complex into the respective protein antigens. The recombinant vaccine is optimized for immunogenicity and enables presentation of diverse antigenic epitopes on both HLA-class I as well as HLA-class II molecules. Consecutively, antigen-specific CD8+ and CD4+ T cell responses will be triggered by HLA-peptide complexes on the surface of antigen presenting cells. In addition, RNA administration will also lead to transient activation (change of surface marker expression and cytokine secretion) of APCs in the targeted lymph nodes particularly via signaling of TLR 7 and 8 leading to an adjuvant effect, supporting the induction of target-specific T cell responses with systemic anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIC, IIIA-C or unresectable stage IV of cutaneous melanoma (AJCC 2009 melanoma classification)
* First line therapy for subjects not eligible or declining other first line therapies after all available treatment options have been transparently disclosed (to be documented!)
* Antigen expression confirmed by RT-PCR analysis from FFPE
* ≥ 18 years of age
* Written informed consent (part I and part II)
* ECOG performance status (PS) 0-1 or Karnofsky Index 70-100 %
* Life expectancy > 3 months
* WBC ≥ 3x109/L
* Hemoglobin ≥ 10 g/dl
* Platelet count ≥ 100,000/mm³
* LDH level < 2.0 x ULN
* Negative pregnancy test (measured by β-HCG) for females of childbearing age
* Suitable lymph nodes for injection using ultrasound guidance

Exclusion Criteria:

* Pregnancy or breastfeeding
* Primary ocular melanoma
* Presence of history (< 5 years) of a second malignancy other than squamous or basal cell carcinoma, non-active prostate cancer or cervical carcinoma in situ
* Brain metastases
* Known or symptomatic pleural effusions and/or ascites
* Known hypersensitivity to the active substance or to any of the excipients
* A serious local infection (e. g. cellulitis, abscess) or systemic infection (e. g. pneumonia, septicemia) which requires systemic antibiotic treatment within 2 weeks prior to the first dose of study medication
* Acute or chronic active hepatitis B or C infection, EBV or CMV
* Receipt of allogenic stem cell transplantation
* Clinically relevant autoimmune disease
* Systemic immune suppression:
* HIV disease
* Use of chronic oral or systemic steroid medication (topical or inhalational steroids are permitted) Other clinical relevant systemic immune suppression
* Symptomatic congestive heart failure (NYHA 3 or 4)
* Unstable angina pectoris
* Radiotherapy, chemotherapy, major surgery, immunotherapy, vaccination, any other concurrent anticancer therapy or any investigational drug within 28 days before the first treatment of this study
* Minor surgery within 14 days before the first treatment of this study
* Treatment with Ipilimumab within 84 days before the first treatment of this study
* Fertile males and females who are unwilling to employ adequate means of contraception (e. g. condom with spermicide, diaphragm with spermicide, birth control pills, injections, patches or intrauterine device) during study treatment and 28 days after the last dose of study treatment
* Presence of a serious concurrent illness or other condition (e. g. psychological, family, sociological, or geographical circumstances) that does not permit adequate follow-up and compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 90 days
  Number of Patients with adverse events, total number of adverse events, dose-limiting toxicities

SECONDARY OUTCOMES:
Determination of antitumoral immune responses | 90 days
  Cellular immune responses, cytokines, AB responses, serum biomarkers, and further immunological parameters will be determined once or repeatedly in the course of treatment. In the latter case changes from baseline will be tabulated.
Clinical Monitoring of Tumor Lesions | 90 days
  Tumor lesion status as determined by CT or MRI results evaluated by irRC and RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Sahin, Prof. Dr., Study Director — Ribological GmbH
Locations (4):
- Medizinische Universität Wien, Abteilung für Dermatologie, Vienna, Austria
- Germany (3):
  - Medizinische Fakultät der Universität Duisburg-Essen, Essen
  - Universtitätsmedizin der Johannes-Gutenberg Universtität, Mainz
  - Universitätsklinik Mannheim, Mannheim